CLINICAL TRIAL: NCT00291967
Title: Evaluate the Feasibility of GSK Biologicals' Tritanrix™-HepB/Hib-MenAC Vaccine Administered as a 3 Dose Primary Vaccination Course at 6, 10 & 14 Weeks of Age
Brief Title: Assess Immune Response Following Primary Vaccination With Tritanrix™-HepB Vaccine Mixed With 3 Formulations of Hib-MenAC Vaccine to Infants
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 759346
Record Dates: First submitted 2006-02-14; First posted 2006-02-15 (Estimated); Last update posted 2006-12-08 (Estimated); Status verified 2006-12

CONDITIONS: Diphtheria; Tetanus; Pertussis; Hepatitis B; Hib Diseases; Neisseria Meningitidis Serogroups A & C Diseases
MeSH Terms: conditions — Diphtheria; Tetanus; Whooping Cough; Hepatitis B

INTERVENTIONS:
Biological: DTPw-HBV/Hib-MenAC conjugate vaccine

SUMMARY:
To compare three formulations of Hib-MenAC vaccines mixed with Tritanrix™-HepB vaccine with that of Tritanrix™-HepB vaccine concomitantly administered with GSK Biologicals' Hiberix™ vaccine and Tritanrix™-HepB vaccine mixed with Hiberix™ vaccine and concomitantly administered with Wyeth Lederle's meningococcal C conjugate vaccine (Meningitec™), with respect to antibody response to vaccine antigens (meningococcal serogroups A and C and PRP) after a three-dose primary vaccination course.

DETAILED DESCRIPTION:
Randomized study with five groups to receive one of the following vaccination regimens: One of the three formulations of GSK Biologicals' Hib-MenAC mixed with GSK Biologicals' Tritanrix™-HepB (3 different groups) GSK Biologicals' Tritanrix™-HepB + GSK Biologicals' Hiberix™ GSK Biologicals' Tritanrix™-HepB mixed with GSK Biologicals' Hiberix™ + Wyeth Lederle's Meningitec™

ELIGIBILITY:
Inclusion Criteria:

* Healthy infant between 6 and 10 weeks of age at the time of the first vaccination, written informed consent obtained from the parents, born after a gestation period of 36 to 42 weeks.

Exclusion criteria:

* Use of any investigational or non-registered product (drug or vaccine) other than the study vaccine(s) or planned administration/ administration of vaccine not foreseen by the study protocol within 30 days preceding the first dose of study vaccine during study period, or planned use during study period with exception of oral polio vaccine (OPV).
* Chronic administration of immunosuppressants or other immune-modifying drugs since birth.
* Hepatitis B and Bacille Calmette-Guérin (BCG) vaccine received after the first 2 weeks of life.
* Any confirmed or suspected immunosuppressive or immunodeficient condition based on medical history and physical examination.
* Administration of immunoglobulins and/or any blood products since birth or planned administration during the study period.
* Previous vaccination against diphtheria, tetanus, pertussis, hepatitis B, Haemophilus influenzae type b, and/or meningococcal disease with the exception of a birth dose of hepatitis B vaccine.

Ages: 6 Weeks to 10 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 525
Dates: Start 2002-11

PRIMARY OUTCOMES:
One month after the third dose of the primary vaccination course, measurement of serum bactericidal titers against meningococcal serogroups A and C (SBA-MenA; SBA-MenC) and anti-PRP antibody concentration.

SECONDARY OUTCOMES:
Immunogenicity: Before the first dose, antibody concentrations or titres against vaccine antigens (MenA, MenC, PRP, pertussis)
One month after the third dose, antibody concentrations or titres against all vaccine antigens
Reactogenicity & safety: after each dose: solicited (d 0-7, local & general) & unsolicited (d 0-30) symptoms
Over the full course of the study: serious adverse events (SAEs)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- Manila, Philippines